CLINICAL TRIAL: NCT05899803
Title: The Effect of the Use of a Walker in Infancy on the Musculoskeletal System and the Level of Physical Activity
Brief Title: Use of Walkers in Infancy and Musculoskeletal System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozden Gokcek (Other)
Responsible Party: Sponsor-Investigator, Ozden Gokcek, Principal Investigator, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023/23
Record Dates: First submitted 2023-05-23; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Use of a Walker in Infancy; Physical Activity Level; Musculoskeletal Problems
Keywords: Baby equipment; physical activity; muscle strength; posture; walker
MeSH Terms: conditions — Motor Activity | interventions — Muscle Strength

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using Walker Group (Experimental): Children who used baby walkers during childhood were included in this group. All assessment procedures were then performed.
  Interventions: Diagnostic Test: Posture Analysis; Diagnostic Test: Physical activity level; Diagnostic Test: Muscle strength
- Walker-Free Group (Active Comparator): Children who did not use a baby walker during childhood were included in this group. All assessment procedures were then performed.
  Interventions: Diagnostic Test: Posture Analysis; Diagnostic Test: Physical activity level; Diagnostic Test: Muscle strength

INTERVENTIONS:
Diagnostic Test: Posture Analysis — This analysis consists of 13 different body parts and evaluates the body in terms of current posture changes. Our study evaluated children from two angles: posterior (head, shoulders, back, hips, feet, and arches) and lateral (neck, chest, shoulders, upper back, trunk, abdomen, and waist). In the scoring system, correct posture was recorded as five points, a moderate amount of deformity posture as three points, and severe deformity posture as one point. The total score calculated at the end of the questionnaire was a maximum of 65 points and a minimum of 13 points. The results of the analysis were evaluated as follows: ≥ 45 points, very good, 40-44 points good, 30-39 points moderate, 20-29 points poor, and a total score of ≤ 19 points.
  Other Names: New York Posture Analysis
Diagnostic Test: Physical activity level — This questionnaire, administered to children aged 4-14, evaluates the activities performed during a week. The questionnaire consisted of nine questions, each of which was evaluated on a 5 points. One point indicated a low physical activity level and five points indicated a high physical activity level. Dividing the total score of the selected items by the number of items gives a summary score for the PAQ-C questionnaire. In our study, we used the Turkish version of the questionnaire, which was found to be reliable and valid.
  Other Names: Physical Activity Questionnaire for Children (PAQ-C)
Diagnostic Test: Muscle strength — Our study objectively measured muscle strength using the JTech Commander PowerTrack Muscle Dynamometer.
  Right and left muscle tests: Hip flexors/hyperextensors/adductors/abductors/internal rotators/external retractors, knee flexors/extensors, and foot plantar flexors/dorsiflexors were evaluated. The measurement results were recorded in Newtons, the measurements were repeated three times, and the average of these three repetitions was recorded.
  Other Names: Digital Muscle Strength Meter

SUMMARY:
The aim of this study was to compare lower extremity muscle strength, posture disorders and physical activity levels of children with and without walker use during infancy. Thirty-nine children aged between 8 and 15 years were included. Demographic data, New York Posture Analysis Questionnaire and Physical Activity Assessment Questionnaire Scale (PAQ-C) were collected. Muscle strength was measured with a digital muscle strength meter.

DETAILED DESCRIPTION:
This study aimed to compare lower extremity muscle strength, postural disorders, and physical activity levels of children who used and did not use a walker during infancy.

The study included 39 children aged between 8 and 15 years. The demographic information of the children, their motor development stages and walker use situations, the age at which they started using it, and the duration of use were questioned. The New York Posture Analysis Questionnaire and Physical Activity Assessment Questionnaire Scale (PAQ-C) were administered to the children. Muscle strength was measured with a digital muscle strength meter.

ELIGIBILITY:
Inclusion Criteria:

* No idiopathic serious orthopedic problems
* No chronic disease
* Children and their parents who volunteered to participate in the study

Exclusion Criteria:

* Presence of neurologic disease.
* Presence of neuromuscular disease.
* Presence of mental retardation.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 6 months
  JTech Commander PowerTrack Muscle Dynamometer
Physical activity level | 6 months
  Physical Activity Questionnaire for Children (PAQ-C)

SECONDARY OUTCOMES:
Posture analysis | 6 months
  New York Posture Analysis Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ege university faculty of health sciences, Izmir, Karsıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
When deemed appropriate, data can be requested from the corresponding author via e-mail.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It can be requested within a period of two years from the year of publication of the work.
Access Criteria: If the data are necessary for the conduct or conclusion of another study, they may be requested from the author.